CLINICAL TRIAL: NCT01695577
Title: Vestibular Rehabilitation and Balance Training for Patients With Dizziness and Balance Problems After Traumatic Brain Injury.
Brief Title: Vestibular Rehabilitation and Balance Training After Traumatic Brain Injury
Acronym: VRTBI2012
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo University College (Other)
Responsible Party: Principal Investigator, Ingerid Kleffelgård, Physical Therapist/ PhD student, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OUSHIOA2012; 2012/195b (Other: REK); 2012/1623 (Other: Personvernombudet OUS)
Record Dates: First submitted 2012-09-19; First posted 2012-09-28 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Traumatic Brain Injury; Brain Concussion; Head Injury; Dizziness
Keywords: Traumatic brain injury; Dizziness; Vestibular rehabilitation; Balance rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Craniocerebral Trauma; Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multidisciplinary evaluation and VR (Experimental): Vestibular rehabilitation and balance training. Twice a week for eight weeks.Outcome measures and tests at baseline, after 8 weeks and 6 months after the injury.
  Interventions: Other: Multidisciplinary evaluation and VR
- Multidisciplinary evaluation and no VR (Active Comparator): Multidisciplinary evaluation. Outcome measures and tests at baseline, after 8 weeks and 6 months after the injury.
  Interventions: Other: Multidisciplinary evaluation

INTERVENTIONS:
Other: Multidisciplinary evaluation and VR — Multidisciplinary assessment and evaluation and VR - Vestibular rehabilitation and balance training. Individually adjusted exercises in groups twice a week for two months. Home exercise program.
  Other Names: Multidisciplinary evaluation and Vestibular rehabilitation
  Arms: Multidisciplinary evaluation and VR
Other: Multidisciplinary evaluation — Multidisciplinary assessment and evaluation.
  Other Names: Multidisciplinary assessment and evaluation.
  Arms: Multidisciplinary evaluation and no VR

SUMMARY:
The main aim of this study is to evaluate the effect of vestibular rehabilitation and balance training on patients with dizziness and balance problems after traumatic brain injury.

DETAILED DESCRIPTION:
8 000 to 10 000 persons are admitted to hospitals in Norway with traumatic brain injury (TBI)annually. Dizziness and balance problems have an incidence of 30-80% in this population.

Studies show that dizziness and imbalance has the potential to restrict several aspects of personal and social life.

Vestibular rehabilitation (VR) is an accepted and effective treatment for dizziness and imbalance. However there is lack of evidence/knowledge about its effect on TBI patients.

The study is designed as a randomized controlled trial study (RCT). Patients aged 16-60 admitted to Oslo University Hospital with TBI and symptoms of dizziness and imbalance are included 8 weeks after the injury.

The intervention and control group will receive multidisciplinary assessment and evaluation. The intervention group will in addition receive group training and a home exercise program by physiotherapists. The intervention will consist of a individually adapted Vestibular Rehabilitation and balance program.

The main outcome measurement is the Dizziness Handicap Inventory (DHI). The study has several other self-report and performance based outcome measures. The outcome measures will be performed before and after the intervention and 6 months after the injury.

ELIGIBILITY:
Inclusion Criteria:

* TBI patients enrolled at Oslo University Hospital.
* persistent dizziness and/or balance problems 2 months post-injury.
* functionally and cognitively able to attend a group training program with vestibular rehabilitation and balance training as the main focus.

Exclusion Criteria:

* severe psychiatric disorder,
* language problems,
* cognitive dysfunction that makes self-report difficult,
* extremity injuries,
* not being able to walk.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | Up to 12 months post injury
  The Dizziness Handicap Inventory (DHI) was developed to measure the self-perceived level of handicap associated with the symptom of dizziness (Jacobson, 1990). The DHI is a 25 item self-report questionnaire with 3 response levels: yes = 4, sometimes = 2, no = 0. The total score is obtained by summing the ordinal scale responses obtained from the 3 response levels (0-100, higher score indicates worse handicap) (Jacobson, 1990).
  The DHI has been translated into Norwegian and has demonstrated satisfactory measurement properties (Tamber, 2009).

SECONDARY OUTCOMES:
High level mobility assessment tool for traumatic brain injury (HiMAT) | Up to 12 months post injury
  The HiMAT is a uni-dimensional performance-based measure of balance and mobility. It consists of 13 walking, running, skipping, hopping and stair items that are measured either by a stopwatch or tape-measure. Raw scores measured in times and distances are noted and converted to a score on a 5-point scale from 0-4, except the two dependent stair items that are rated on a 6- point scale from 0-5. A 0 corresponds to inability to perform the item, and 1 -4/5 represents increasing levels of ability. The sum score range is 0-54 (worst-best). A user/instruction manual for the testers describing the test in detail is developed. (Williams, 2006;Williams, 2006).

OTHER OUTCOMES:
Balance Error Scoring System (BESS). | Up to 12 months post injury
  The Bess is a standardized balance testing system. It consists of three 20 second, standardized stances on a firm surface and on a foam surface with eyes closed. The stances are: double leg stance, single-leg stance and tandem stance. Errors are counted during each 20-second trial(Bell, 2011;Finnoff, 2009). The Bess has variable but satisfactory measurement properties and norms are developed (Bell, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Ingerid Kleffelgård, MSc., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided